CLINICAL TRIAL: NCT03996538
Title: Vaccination Efficacy With Metformin in Older Adults: A Pilot Study
Brief Title: Vaccination Efficacy With Metformin in Older Adults
Acronym: VEME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Jenna Bartley, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-205-2; 18155 (Other Grant/Funding Number: AFAR)
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Aging; Age-Related Immunodeficiency; Vaccine Response Impaired
MeSH Terms: interventions — Metformin; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Metformin and placebo tablets will be identical. Participants and researchers will not know treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin Hydrochloride Extended Release Tablets (Experimental): Patients will consume 3 tablets of 500mg metformin hydrochloride extended-release tablets daily (1500mg/day (after 3 week dose gradation)).
  Interventions: Drug: Metformin Hydrochloride Extended-Release Tablets; Biological: Influenza Vaccine
- Placebo (Placebo Comparator): Patients will consume 3 identical placebo tablets (after similar 3 week dose gradation).
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Drug: Metformin Hydrochloride Extended-Release Tablets — Subjects will ingest 1500mg/day of metformin hydrochloride extended release. Immune responses will be examined prior to treatment, prior to flu vaccination, and after flu vaccination.
  Other Names: metformin hydrochloride ER; metformin hcl ER; metformin ER
  Arms: Metformin Hydrochloride Extended Release Tablets
Biological: Influenza Vaccine — All subjects will be vaccinated with high-dose influenza vaccine at the appropriate time of the year per current CDC and FDA recommendations
  Other Names: Flu Vaccine

SUMMARY:
With aging the immune system gets weaker. This makes older adults more susceptible to influenza (flu). Vaccinations help to prevent infection from the flu virus, however the immune system of older adults do not respond as well to vaccines compared to young adults and thus, aren't as well protected from the complications from the flu. This research is being done to determine if Metformin, an FDA-approved diabetes medication, is effective at enhancing immune responses to flu vaccine in older men and women. Participants will be randomly assigned to either metformin or placebo treatment for a total of 22 weeks. Participants will be vaccinated with high-dose flu vaccine after 12 weeks of treatment. Immune responses will be evaluated throughout the study at 6 time points.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 65 years and older
* Willingness to provide consent and participate in all aspects of the trial including randomization to the intervention group and receiving this year's flu vaccine
* Received previous year's seasonal influenza vaccine

Exclusion Criteria:

* History of severe renal impairment and/or eGFR ≤ 45 mL/min/1.73m2
* Excessive alcohol use (more than 14 alcoholic drinks/week) or clinical/laboratory evidence of hepatic disease (via medical history and/or AST and/or ALT ≥ 3 times upper limit of normal at screening)
* Acute or chronic metabolic acidosis (via medical history and/or low serum bicarbonate (< 22mEq/L), increased anion gap (> 10 mEq/L))
* History of B12 deficiency within the last 10 years
* Known type 2 diabetes or screening of prediabetic (HbA1c 5.7-6.4%) or diabetic (HbA1c ≥ 6.5%)
* Currently taking metformin or other diabetes medications
* Unwilling or unable (due to significant cognitive impairment) to provide informed consent
* Terminal illness with life expectancy less than 12 months
* Advanced neurological disorder (Parkinson's, ALS, MS, dementia)
* Cancer or history of cancer in the past 2 years (excluding non-melanoma skin cancer) or any history of metastatic (stage 4) cancer
* Significant co-morbid disease (severe chronic obstructive pulmonary disease, active rheumatologic diseases, chronic infection (HIV, tuberculosis), severe congestive heart failure (NYHA class 4), myocarditis, etc)
* Myocardial infarction, stroke or hospitalization for heart failure in the last 12 months
* Severe active psychiatric disorder (e.g. bipolar, schizophrenia)
* Unable to complete physical performance testing due to medical conditions (at discretion of the PI)
* Uncontrolled hypertension (systolic/diastolic blood pressure >150/90 mmHg)
* Unintentional weight loss >10% in past 12 months
* Allergy or history of adverse reaction to flu vaccine or any ingredients in flu vaccine, including eggs
* History of Guillain-Barre syndrome following vaccination
* Immunosuppressive disorders or taking immunosuppressive medications (including oral prednisone > 10mg/day)
* Current participation in another interventional study
* Refusal to receive flu vaccine

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Change in Cell-mediated Flu Vaccine Responses - inducible Granzyme B | Prior to vaccination (week 12) and 5 weeks post vaccination (week 17)
  Change in inducible Granzyme B levels in peripheral blood mononuclear cells (PBMCs) stimulated ex vivo with live flu virus will be compared between the metformin and placebo group.
Change in Cell-mediated Flu Vaccine Responses - interferon(IFN)-γ/interleukin(IL)-10 ratio | Prior to vaccination (week 12) and 5 weeks post vaccination (week 17)
  Change in interferon(IFN)-γ/interleukin(IL)-10 ratio in culture supernatant of peripheral blood mononuclear cells (PBMCs) stimulated ex vivo with live flu virus will be compared between the metformin and placebo group.

SECONDARY OUTCOMES:
Change in Influenza Antibody Titers | Prior to treatment (week 0), prior to vaccination (week 12), and after vaccination (week 13, 17, and 22)
  Serum antibody titers will be analyzed via hemagglutination inhibition assays (HI) via established Center for Disease Control (CDC) and World Health Organization (WHO) protocols for each vaccine strain. Change in antibody titer levels over time will be evaluated.
Change in T Cell Metabolic Phenotype | Prior to treatment (week 0), prior to vaccination (week 12), and after vaccination (week 13, 17, and 22)
  T cells will be evaluated for phenotypic differences of glucose transporter expression via flow cytometry and reported as percent positive cells. Change in percent positive cells over time will be evaluated.
Change in T Cell Oxygen Consumption Rate | Prior to treatment (week 0), prior to vaccination (week 12), and after vaccination (week 13, 17, and 22)
  T cells will be evaluated for oxygen consumption rate via Seahorse Agilent Technologies. Change in oxygen consumption rate over time will be evaluated.
Change in Frailty Phenotype | Prior to treatment (week 0), prior to vaccination (week 12), and after vaccination (week 13, 17, and 22)
  Subjects will complete frailty testing via Fried Frailty Phenotype. Change in frailty phenotype over time will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna M Bartley, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States